CLINICAL TRIAL: NCT02548286
Title: A Randomized, Open-label, Single-dosing, Crossover Study to Compare the Safety and Pharmacokinetics of CKD-330(Fixed-dose Combination of Candesartan Cilexetil 8 mg and Amlodipine 5 mg) With Coadministration of the Two Separate Drugs in Healthy Male Volunteers(B)
Brief Title: Study to Compare the Safety and Pharmacokinetics of CKD-330 8/5mg With Coadministration of the Two Separate Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 144BE15015
Record Dates: First submitted 2015-08-20; First posted 2015-09-14 (Estimated); Last update posted 2015-12-07 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: Hypertension; Healthy male volunteer; Candesartan, Amlodipine
MeSH Terms: conditions — Hypertension | interventions — candesartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Candesartan and Amlodipine (Active Comparator): Candesartan 8mg and Amlodipine 5mg, PO, 1day or 22day
  Interventions: Drug: Candesartan 8mg; Drug: Amlodipine 5mg
- CKD-330 (Experimental): CKD-330 8/5mg, PO, 1day or 22day
  Interventions: Drug: CKD-330 8/5mg

INTERVENTIONS:
Drug: Candesartan 8mg — PO, 1day or 22day
  Arms: Candesartan and Amlodipine
Drug: Amlodipine 5mg — PO, 1day or 22day
  Arms: Candesartan and Amlodipine
Drug: CKD-330 8/5mg — PO, 1day or 22day
  Arms: CKD-330

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetics of CKD-330 (fixed-dose combination of Candesartan Cilexetil 8 mg and Amlodipine 5 mg) with coadministration of the two separate drugs in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteer in the age of 19-45
2. Body weight ≥ 55 kg and in the range of calculated IBW ±20%
3. Subject without a hereditary problems, chronic disease and morbid symptom
4. Suitable clinical laboratory test values
5. Subject who sign on an informed consent form willingly

Exclusion Criteria:

1. Clinically significant disease with hepatobiliary, nephrological, neurologic, respiratory, haemato-oncological, endocrine, urogenital, psychiatric, musculoskeletal, immune, otorhinolaryngological, cardiovascular system
2. Gastrointestinal disease or gastrointestinal surgery
3. History of significant hypersensitivity reaction of amlodipine, candesartan, calcium channel blocker, angiotensin II receptor blocker or other drugs
4. Galactose intolerance
5. Sitting systolic blood pressure ≥ 140 mmHg or< 90 mmHg, sitting diastolic blood pressure ≥ 95 mmHg or < 60 mmHg, pulse ≥ 100 beats per minute
6. Aspartate aminotransferase, Alanine aminotransferase, Total bilirubin > 2 x upper limit of normal range
7. Serum Creatinine > upper limit of normal range
8. Drug abuse
9. Subject treated metabolizing enzyme inducers or inhibitors within 1 month
10. Subject treated ethical the counter or herbal medicine within 2 weeks, over-the-counter or vitamin within 1 week
11. Subject treated Investigational product(include Bioequivalence test) within 3 months
12. Whole blood donation within 2 months, component blood donation or blood transfusion within 1 month
13. Continuously taking Alcohol > 21 units/week
14. Cigarette > 10 cigarettes/day
15. Subjects with planning of dental treatment or any surgery
16. Another clinical condition in judgement of investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Cmax(Maximum Plasma Concentration) of Candesartan | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
AUCt(Area Under the Plasma Concentration-time curve) of Candesartan | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
Cmax(Maximum Plasma Concentration) of Amlodipine | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
AUCt(Area Under the Plasma Concentration-time curve) of Amlodipine | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr

SECONDARY OUTCOMES:
AUCinf(Area Under the Plasma Concentration-time curve from time t to infinity) of Candesartan | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
tmax(Time to reach the maximum concentration) of Candesartan | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
t1/2β(Time for C max to drop in half) of Candesartan | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
CL/F(Clearance/Bioavailability) of Candesartan | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48 hr
AUCinf(Area Under the Plasma Concentration-time curve from time t to infinity) of Amlodipine | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
tmax(Time to reach the maximum concentration) of Amlodipine | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
t1/2β(Time for C max to drop in half) of Amlodipine | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr
CL/F(Clearance/Bioavailability) of Amlodipine | 0(Pre-dose), 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hr

CONTACTS AND LOCATIONS:
Overall Officials: Jang Hee Hong, MD, PhD, Principal Investigator — Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, Jung-gu, South Korea